CLINICAL TRIAL: NCT06859619
Title: Seroprevalence of Zoonotic and Arboviral Emerging Infections in Exposed Agents from the City of Montpellier: a Transversal Study.
Brief Title: Serological Measurement of Montpellier Professionals' Contacts with Infectious Agents Responsible for Animal-borne Diseases
Acronym: SEZAM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: TransVIHMI UM, IRD UMI233, Inserm U1175 (Unknown); UMR 1058 Pathogenesis & Control of Chronic & Emerging Infections PCCEI (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: RECHMPL24_0384
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Leishmaniasis; Leptospirosis; Brucellosis; Q Fever; Rickettsiosis; Tularemia; Psittacosis; Lyme Disease; Tick-borne Encephalitis; Hantaviral Infection Nos; Hepatitis E; Dengue Virus; Zika Virus; Chikungunya Virus Infection; West Nile Virus; Usutu Virus; Toscana Virus; Crimean-Congo Haemorrhagic Fever Virus
Keywords: Leishmaniasis,; Leptospirosis; Brucellosis; Zika virus; Q fever, Rickettsiosis; Lyme disease; Tick-borne encephaliti; Hantavirus; Hepatitis E virus; Dengue virus; Chikungunya virus; West-Nile virus; Usutu virus; Toscana virus; Tularemia; Psittacosis; Crimean-Congo haemorrhagic fever virus; epidemiology
MeSH Terms: conditions — Leishmaniasis; Leptospirosis; Brucellosis; Q Fever; Rickettsia Infections; Tularemia; Psittacosis; Lyme Disease; Encephalitis, Tick-Borne; Hepatitis E; Zika Virus Infection; Chikungunya Fever; Hantavirus Pulmonary Syndrome

STUDY DESIGN:
Intervention Model Description: cross-sectional study with minimal risk and constraints
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- City of Montpellier employees working at the Zoo, the Ecolothèque and the Green Spaces Department (Experimental): City of Montpellier employees working at the Zoo, Ecolotheque or green spaces exposed to wildlife by zoo staff and to various vectors (ticks, mosquitoes, sandflies) in the Occitanie region
  Interventions: Other: Peripheral venous blood sample

INTERVENTIONS:
Other: Peripheral venous blood sample — Peripheral venous blood sampling for IgG serology against leishmaniasis, leptospirosis, brucellosis, Q fever, rickettsiosis, tularemia, psittacosis, Lyme disease, tick-borne encephalitis, hantavirus, hepatitis E virus, dengue virus, Zika virus, Chikungunya virus, West Nile virus, Usutu virus, Toscana virus, Crimean-Congo hemorrhagic fever virus.

SUMMARY:
Zoonoses and arboviroses refer to a group of diseases transmitted from animals to humans, either directly or indirectly (via mosquitoes, ticks or contact with contaminated environments). Most of these diseases are found in certain tropical zones, but global warming and increased international trade are modifying their geographical distribution, with a gradual trend towards temperate regions. A number of these pathogens have already been detected in Occitania, including dengue fever, West Nile, leishmaniasis and Q fever. Given the region's high mosquito population and favorable climatic conditions, other zoonoses have a strong potential to appear in the region, or may already be circulating at a low level. The study focuses on 18 pathogens selected for their potential to emerge and establish themselves in the Occitanie region: Leishmaniasis, Leptospirosis, Brucellosis, Q fever, Rickettsiosis, Tularemia, Psittacosis, Lyme disease, Tick-borne encephalitis, Hantavirus, Hepatitis E virus, Dengue virus, Zika virus, Chikungunya virus, West-Nile virus, Usutu virus, Toscana virus, Crimean-Congo haemorrhagic fever virus.

The aim of the study is to find out whether patients have antibodies against these infectious agents, which would indicate that they have been exposed to them in the past, even in the absence of symptoms.

Describing the circulation of these pathogens will enable to implement appropriate public health measures to avoid the risk of epidemics (mosquito control, informing professionals, etc.), as well as to assess the risk incurred in the workplace and have this risk recognized by the healthcare system.

DETAILED DESCRIPTION:
Current environmental changes are influencing the epidemiology of zoonoses, which account for over 75% of emerging infections, with the Mediterranean region being a high-risk area. The proposed study focuses on occupational zoonoses, that is, those that can be contracted in the workplace, through direct contact with animals or exposure to their environment. Some of these zoonoses are recognized and compensable as occupational diseases (OD), while for others, the onus is on the employee to prove the origin of the contamination. The advantages of studying this population are threefold: i) to document occupational risk and improve management and prevention practices in this context, ii) to use this sentinel population - when many of these zoonoses are emerging - to anticipate risks for the less-exposed general population, iii) in the event of the discovery of a positive serology for an infectious agent considered non-circulating in the Occitanie region, to improve the management of symptomatic patients by raising awareness of differential diagnosis. For the purposes of this study, the zoonoses recognized as occupational diseases are: Mediterranean spotted fever, Lyme borreliosis, tularemia, Q fever, brucellosis, psittacosis, hepatitis E and leptospirosis. Although not recognized as occupational diseases, leishmaniasis, hantaviruses, dengue fever, zika, chikungunya, West Nile virus, Usutu, Toscana, Crimean-Congo hemorrhagic fever and tick-borne encephalitis are of particular interest to workers exposed to these diseases, and are also included in the study.

Few data are currently available on the actual rate of circulation of these pathogens in the population of occupationally exposed workers, and none in Occitanie. These outdoor workers also represent a sentinel population, due to their increased exposure, so obtaining precise seroprevalence data in these groups would enable the researchers to anticipate the emergence of these pathogens in the general population in the near future, and to diagnose them individually.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Consultant in an infectious diseases department
* Have given written consent to participate in the study
* Working for the City or Metropolis of Montpellier in the Zoo, Espaces Vert or Ecolothèque departments.

Exclusion Criteria:

* - Pregnant and breast-feeding women
* Persons benefiting from legal protection measures (guardianship, curatorship, safeguard of justice)
* Participants who are not fluent in French and who do not have a support person capable of reading French.
* Persons unable to express their consent.
* Persons participating in another research project with an exclusion period still in progress.
* Persons not affiliated to a social security scheme or not benefiting from such a scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Estimated)
Dates: Start 2025-03-03 (Estimated); Primary Completion 2025-10-03 (Estimated); Study Completion 2025-10-03 (Estimated)

PRIMARY OUTCOMES:
Estimate seroprevalences of the zoonoses in populations exposed to wildlife by zoo staff and to various vectors (ticks, mosquitoes, sandflies). Leishmaniasis, | Baseline
  prevalence (in percentage) of pathogen IgG positivity against : Leishmaniasis,
Estimate seroprevalences of the zoonoses in populations exposed to wildlife by zoo staff and to various vectors (ticks, mosquitoes, sandflies).Leptospirosis, | Baseline
  prevalence of pathogen IgG positivity against : Leptospirosis,
Estimate seroprevalences of the zoonoses in populations exposed to wildlife by zoo staff and to various vectors (ticks, mosquitoes, sandflies).Brucellosis | Baseline
  prevalence of pathogen IgG positivity against : Brucellosis
Estimate seroprevalences of the zoonoses in populations exposed to wildlife by zoo staff and to various vectors (ticks, mosquitoes, sandflies).Q fever | Baseline
  prevalence of pathogen IgG positivity against : Q fever
Estimate seroprevalences of the zoonoses in populations exposed to wildlife by zoo staff and to various vectors (ticks, mosquitoes, sandflies).Rickettsiosis | Baseline
  prevalence of pathogen IgG positivity against : Rickettsiosis,
Estimate seroprevalences of the zoonoses in populations exposed to wildlife by zoo staff and to various vectors (ticks, mosquitoes, sandflies).Tularemia | Baseline
  prevalence of pathogen IgG positivity against : Tularemia
Estimate seroprevalences of the zoonoses in populations exposed to wildlife by zoo staff and to various vectors (ticks, mosquitoes, sandflies).Psittacosis | Baseline
  prevalence of pathogen IgG positivity against : Psittacosis
Estimate seroprevalences of the zoonoses in populations exposed to wildlife by zoo staff and to various vectors (ticks, mosquitoes, sandflies).Lyme disease, | Baseline
  prevalence of pathogen IgG positivity against : Lyme disease,
Estimate seroprevalences of the zoonoses in populations exposed to wildlife by zoo staff and to various vectors (ticks, mosquitoes, sandflies).Tick-borne encephalitis | Baseline
  prevalence of pathogen IgG positivity against : Tick-borne encephalitis
Estimate seroprevalences of the zoonoses in populations exposed to wildlife by zoo staff and to various vectors (ticks, mosquitoes, sandflies).Hantavirus | Baseline
  prevalence of pathogen IgG positivity against : Hantavirus
Estimate seroprevalences of the zoonoses in populations exposed to wildlife by zoo staff and to various vectors (ticks, mosquitoes, sandflies). Hepatitis E virus | Baseline
  prevalence of pathogen IgG positivity against : Hepatitis E virus
Estimate seroprevalences of the zoonoses in populations exposed to wildlife by zoo staff and to various vectors (ticks, mosquitoes, sandflies).Dengue virus | Baseline
  prevalence of pathogen IgG positivity against : Dengue virus
Estimate seroprevalences of the zoonoses in populations exposed to wildlife by zoo staff and to various vectors (ticks, mosquitoes, sandflies). Zika virus | Baseline
  prevalence of pathogen IgG positivity against : Zika virus
Estimate seroprevalences of the zoonoses in populations exposed to wildlife by zoo staff and to various vectors (ticks, mosquitoes, sandflies).Chikungunya virus | Baseline
  prevalence of pathogen IgG positivity against : Chikungunya virus
Estimate seroprevalences of the zoonoses in populations exposed to wildlife by zoo staff and to various vectors (ticks, mosquitoes, sandflies). West-Nile virus, | Baseline
  prevalence of pathogen IgG positivity against : West-Nile virus,
Estimate seroprevalences of the zoonoses in populations exposed to wildlife by zoo staff and to various vectors (ticks, mosquitoes, sandflies). usutu virus | Baseline
  prevalence of pathogen IgG positivity against : Usutu virus
Estimate seroprevalences of the zoonoses in populations exposed to wildlife by zoo staff and to various vectors (ticks, mosquitoes, sandflies).Toscana virus | Baseline
  prevalence of pathogen IgG positivity against : Toscana virus
Estimate seroprevalences of the zoonoses in populations exposed to wildlife by zoo staff and to various vectors (ticks, mosquitoes, sandflies).Crimean-Congo haemorrhagic fever virus. | Baseline
  prevalence of pathogen IgG positivity against : Crimean-Congo haemorrhagic fever virus.

SECONDARY OUTCOMES:
Determine the factors associated with seropositivity to these diseases. socio-demographic criteria | Baseline
  OR of logistic regression of univariate model between serologies and socio-demographic criteria (age, sex, profession)
Determine the factors associated with seropositivity to these diseases. travel to endemic areas | Baseline
  OR of the logistic regression of the univariate model between serologies and travel to endemic areas for these diseases
Determine the factors associated with seropositivity to these diseases. occupational exposure | Baseline
  OR of the logistic regression of the univariate model between serologies and occupational exposure to these pathologies
Determine the factors associated with seropositivity to these diseases. exposure in private activities | Baseline
  OR of the logistic regression of the univariate model between serologies and exposure in private activities, including the importance of contact with transmission vectors,
Determine the factors associated with seropositivity to these diseases. use of mosquito protection | Baseline
  OR of the logistic regression of the univariate model between serologies and use of mosquito protection,
Determine the factors associated with seropositivity to these diseases.history of transfusion or transplant | Baseline
  OR of the logistic regression of the univariate model between serologies and history of transfusion or transplant
Determine the factors associated with seropositivity to these diseases. comparison of the linear models | Baseline
  AOR of the multivariate logistic regression with the best AIC among all the models tested
Estimating vaccination coverage against leptospirosis in the workplace | Baseline
  prevalence (in percentage) of professional vaccinations for leptospirosis
Estimating vaccination coverage against rabies in the workplace | Baseline
  prevalence (in percentage) of professional vaccinations for rabies
Determine the sensitivity of DBS (dried blood spot) serum neutralization for viral serologies. Dengue virus | Baseline
  Determine the sensitivity (in percentage) of DBS (dried blood spot) seroneutralization for Dengue virus
Determine the specificity of DBS (dried blood spot) serum neutralization for viral serologies. Dengue virus | Baseline
  Determine the specificity (in percentage) of DBS (dried blood spot) seroneutralization for Dengue virus
Determine the specificity of DBS (dried blood spot) serum neutralization for viral serologies. Zika virus | Baseline
  Determine the specificity (in percentage) of DBS (dried blood spot) seroneutralization for Zika virus
Determine the sensitivity of DBS (dried blood spot) serum neutralization for viral serologies. Zika virus | Baseline
  Determine the sensitivity (in percentage) of DBS (dried blood spot) seroneutralization for Zika virus
Determine the sensitivity of DBS (dried blood spot) serum neutralization for viral serologies. Chikungunya virus | Baseline
  Determine the sensitivity (in percentage) of DBS (dried blood spot) seroneutralization for Chikungunya virus
Determine the specificity of DBS (dried blood spot) serum neutralization for viral serologies. Chikungunya virus | Baseline
  Determine the specificity (in percentage) of DBS (dried blood spot) seroneutralization for Chikungunya virus
Determine the sensitivity of DBS (dried blood spot) serum neutralization for viral serologies. West-Nile virus | Baseline
  Determine the sensitivity (in percentage) of DBS (dried blood spot) seroneutralization for West-Nile virus
Determine the specificity of DBS (dried blood spot) serum neutralization for viral serologies. West-Nile virus | Baseline
  Determine the specificity (in percentage) of DBS (dried blood spot) seroneutralization for West-Nile virus
Determine the sensitivity of DBS (dried blood spot) serum neutralization for viral serologies. Usutu virus | Baseline
  Determine the sensitivity (in percentage) of DBS (dried blood spot) seroneutralization for Usutu virus
Determine the specificity of DBS (dried blood spot) serum neutralization for viral serologies. Usutu virus | Baseline
  Determine the specificity (in percentage) of DBS (dried blood spot) seroneutralization for Usutu virus
Determine the sensitivity of DBS (dried blood spot) serum neutralization for viral serologies. Toscana virus | Baseline
  Determine the sensitivity (in percentage) of DBS (dried blood spot) seroneutralization for Toscana virus
Determine the specificity of DBS (dried blood spot) serum neutralization for viral serologies. Toscana virus | Baseline
  Determine the specificity (in percentage) of DBS (dried blood spot) seroneutralization for Toscana virus
Determine the sensitivity of DBS (dried blood spot) serum neutralization for viral serologies. Crimean-Congo haemorrhagic fever virus | Baseline
  Determine the sensitivity (in percentage) of DBS (dried blood spot) seroneutralization for Crimean-Congo haemorrhagic fever virus
Determine the specificity of DBS (dried blood spot) serum neutralization for viral serologies. Crimean-Congo haemorrhagic fever virus | Baseline
  Determine the specificity (in percentage) of DBS (dried blood spot) seroneutralization for Crimean-Congo haemorrhagic fever virus

CONTACTS AND LOCATIONS:
Overall Officials: CHARLOTTE BOULLE, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital Of Montpellier, Montpellier, herault, France

IPD SHARING:
Plan to Share IPD: Undecided